CLINICAL TRIAL: NCT03869697
Title: A Phase I Study Evaluating the Safety, Tolerability, Efficacy, and Pharmacokinetics of SCB-313, a Fully-Human TRAIL-Trimer Fusion Protein, for the Treatment of Malignant Pleural Effusions
Brief Title: Study With SCB-313 (Recombinant Human TRAIL-Trimer Fusion Protein) for Treatment of Malignant Pleural Effusions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLO-SCB-313-002
Record Dates: First submitted 2019-03-01; First posted 2019-03-11 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Malignant Pleural Effusions
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCB-313 (Experimental): Cohorts in SAD phase: 5 mg, 10mg, 20mg, 40mg, 80 mg. Cohort in MAD phase: biological effective dose determined from SAD phase. 1 intrapleural injection of SCB-313 on Day 1 for the SAD cohorts, and 3 intrapleural injections of SCB-313 on Days 1, 2 and 3 for the MAD cohort.
  Interventions: Drug: SCB-313

INTERVENTIONS:
Drug: SCB-313 — 5 mg or 20 mg lyophilized powder in a single-use glass vial
  Other Names: recombinant human TRAIL-Trimer fusion protein

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, preliminary efficacy, and PK/PD of SCB-313 (recombinant human TRAIL-Trimer fusion protein) administered once via intrapleural injection (SAD) and once daily over 2 to 3 days (MAD)for the treatment of cancer patients with symptomatic malignant pleural effusions requiring drainage.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed cancer of any primary tumor type.
2. Malignant pleural effusion causing respiratory symptoms requiring drainage that is histologically or cytologically confirmed; or pleural effusion with radiologically proven pleural malignancy as diagnosed in normal clinical practice on thoracic computed tomography in the absence of histocytological or cytological proof.
3. Eastern Cooperative Oncology Group (ECOG) performance status: 0 to 2. Patients with an ECOG performance status of 3 may be included if the Investigator determines that removal of pleural fluid would improve their performance status to 2 or better.
4. Life expectancy of at least 8 weeks.
5. Age ≥18 years.
6. Adequate hematologic function, defined as:

   1. Platelet count ≥75,000/μL;
   2. Prothrombin time and activated partial thromboplastin time ≤1.5 times the upper limit of normal (ULN);
   3. Absolute neutrophil count ≥1,500 μL;
   4. Hemoglobin ≥8 g/dL (transfusion and erythropoietic agents are allowed). In case there is existence of active bleeding or other persistent condition of either increased destruction or impaired production of erythrocytes, which may require repeated transfusion or erythropoietic treatment, the eligibility must be discussed with the Sponsor on a case-by-case basis prior to randomization).
7. Adequate renal function, defined as creatinine clearance >40 mL/minute.
8. Adequate liver function, defined as:

   1. Aspartate aminotransferase and alanine aminotransferase ≤2.0 times ULN;
   2. Bilirubin ≤2.0 times ULN, unless patient has known Gilbert's syndrome.
9. Female patients of childbearing potential (excluding women who have undergone surgical sterilization or are menopausal, defined as no menstrual periods for 1 year or more without any other medical reasons) are eligible if they have negative serum pregnancy test result 7 days before the first dose of SCB-313 and are willing to use an effective method of birth control/contraception to prevent pregnancy until 6 months after discontinuation of SCB-313.

   Both men and women of reproductive potential must agree to use effective contraception during the study and for 6 months after discontinuation of SCB-313.

   Note: Contraceptive methods that are considered highly effective areas follows: total abstinence, intrauterine device, double barrier method (such as condom plus diaphragm with spermicide), contraceptive implant, hormonal contraceptives (contraceptive pills, implants, transdermal patches, hormonal vaginal devices, or injections with prolonged release), or vasectomized partner with confirmed azoospermia.
10. Willing to attend follow-up visits on Days 10, and 21 after the first study drug administration.

Exclusion Criteria:

1. Significantly loculated pleural effusions not amenable to drainage or patient is unlikely to benefit from intrapleural therapy.
2. Concurrent use of any investigational product (IP) or investigational medicine within 28 days before Day 1 of study drug administration.
3. Radiotherapy outside the chest field within 2 weeks, or radical radiotherapy to pleural or lung lesions within 8 weeks prior to enrollment (Note: palliative radiotherapy to the chest is allowed).
4. Start a new systemic anticancer therapy, including chemotherapy, targeted therapy, immuno-oncology (I-O) therapy regimen, within 28 days before Day 1 of study drug administration or during DLT observation period.
5. Acute or chronic infection (such as tuberculosis) requiring antiviral or intravenous antibiotics within 2 weeks prior to enrollment.
6. Clinical unstable or uncontrolled concomitant hematologic, cardiovascular, pulmonary, hepatic, renal, pancreatic, or endocrine diseases.
7. History of gross hemoptysis (>2.5 mL).
8. Residual adverse events (AEs) > Grade 2 from previous treatment.
9. Evidence or suspicion of relevant psychiatric impairment, including alcohol or recreational drug abuse.
10. Myocardial infarction within 6 months prior to treatment and/or prior diagnoses of congestive heart failure (New York Heart Association Class III or IV), unstable angina, unstable cardiac arrhythmia requiring medication, and/or long QT syndrome or QT/QTc interval >480 msec at Baseline.
11. Uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg confirmed upon repeated measures (note: no more than 3 repeated measures allowed).
12. Major surgery (open procedures) within 4 weeks prior to enrollment.
13. Patient with ileus within 30 days prior to Screening.
14. Positive serology test for human immunodeficiency virus type 1 and/or 2, or known history of other immunodeficiency disease.
15. Live vaccine within 2 weeks prior to enrollment.
16. Scheduled participation in another clinical study involving an investigational product or device during the DLT observation period of this study.
17. Previous treatment with a TRAIL-based therapy or death receptor 4/5 agonist therapy.
18. Known or suspected hypersensitivity to any component of SCB-313.
19. Any further condition which, in the opinion of the Investigator, may result in undue risk of the patient by participating in the present study.
20. Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Occurrence of DLT | Up to 21 days after start of treatment
  Occurrence of dose limiting toxicity (DLT)

SECONDARY OUTCOMES:
SAEs or TEAEs | Up to 21 days after start of treatment
  Occurrence of serious adverse events (SAEs) and/or treatment-emergent adverse events (TEAEs) regardless of causality or relationship to SCB-313, graded using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03
Immunogenicity | Up to 21 days after start of treatment
  Occurrence of binding and neutralizing anti-SCB-313 antibodies
Pleural effusion response rate at Day 21 | At Day 21 after start of treatment
  Based on chest radiographs at Day 21, compared to Baseline.
Pleural effusion drainage-free rate at Day 21 | At Day 21 after start of treatment
  Defined as the probability of being effusion-drainage free at Day 21
The changes in effusion volume and flow rate after SCB-313 treatment , and at next drainage over the baseline daily effusion flow rate. | Up to 6 months after start of treatment
  1. The baseline daily effusion flow rate will be measured.
  2. Effusion flow rate will be calculated from the effusion volume drained over the time elapsed between drainages.
  3. Effusion flow rate at next pleural drainage will be calculated from the volume over the time elapsed between drainages.
Blood oxygen levels | Up to 21 days after start of treatment
  To compare blood oxygen levels during the study
Overall survival | Up to 6 months after start of treatment
  The time from the first dose of SCB-313 until death from any cause.
Pharmacokinetics (Cmax) | Up to 4 days after start of treatment
  Maximum SCB-313 concentration
Pharmacokinetics(Cmax/D) | Up to 4 days after start of treatment
  Dose-normalized Cmax of SCB-313
Pharmacokinetics(Tmax) | Up to 4 days after start of treatment
  Time to Cmax of SCB-313
Pharmacokinetics ([AUC]0-24) | Up to 4 days after start of treatment
  Area under SCB-313 concentration time curve from zero to 24 hours after dosing
Pharmacokinetics (AUC0-24/D) | Up to 4 days after start of treatment
  Dose-normalized AUC0-24
Pharmacokinetics ((AUC0-last)) | Up to 4 days after start of treatment
  Area under the SCB-313 concentration-time curve from time zero to the last quantifiable concentration time point
Pharmacokinetics (Ctrough) | Up to 4 days after start of treatment
  Trough concentration (Ctrough) at each predose time point and at 24 hours after the last dose
Amount of drug in pleural effusion | Up to 4 days after start of treatment
  Amount of SCB-313 in pleural effusion at 24 hours after each dose
Pharmacokinetics (AUC 0-inf) | Up to 4 days after start of treatment
  Area under the curve from time zero extrapolated to infinity
Pharmacokinetics (AUC0-inf/D) | Up to 4 days after start of treatment
  Dose-normalized AUC0-inf
Pharmacokinetics (t1/2) | Up to 4 days after start of treatment
  Terminal half-life
Pharmacokinetics (CL/F serum only) | Up to 4 days after start of treatment
  Apparent systemic clearance after intrapleural dosing
Pharmacokinetics (Vz/F serum only) | Up to 4 days after start of treatment
  Apparent volume of distribution after intrapleural dosing
Pharmacokinetics (λz) | Up to 4 days after start of treatment
  Terminal rate constant
Tumor response | Up to 6 months after start of treatment
  Tumor response in patients with measurable disease using RECIST v1.1 as applicable.
Carcinoembryonic antigen (CEA) | Up to 21 days after start of treatment
  Changes in serum tumor markers
CA-125 | Up to 21 days after start of treatment
  Changes in serum tumor markers
CA-19-9 | Up to 21 days after start of treatment
  Changes in serum tumor markers
Changes in 24-hour urine volume | Up to 4 days after start of treatment
  Measured urine volume at baseline and postdose
Changes in GFR | Up to 4 days after start of treatment
  The changes in glomerular filtration rate
Changes in tumor cell count in pleural effusion samples | Up to 4 days after start of treatment
  The changes in tumor cell count
Caspase-cleaved CK18 | Up to 10 days after start of treatment
  Changes in serum PD biomarker
KRAS mutation | Baseline
  Predictive biomarker analysis (assessed using archival tumor specimens )
MMR defects | Baseline
  Predictive biomarker analysis (assessed using archival tumor specimens )
Bcl2 overexpression | Baseline
  Predictive biomarker analysis (assessed using archival tumor specimens )
TRAIL resistance | Baseline
  Predictive biomarker analysis (assessed using pleural effusion samples)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Orange Health Service, Orange, New South Wales
  - The Royal Melbourne Hospital, Parkville, Victoria
  - SCGH (Sir Charles Gairdner Hospital), Nedlands, Western Australia